CLINICAL TRIAL: NCT00574431
Title: Implementation of an Evidence-based Nutritional Management Protocol in Critically Ill Patients:Does Clinical Outcome Improve?
Brief Title: ICU Nutrition Study Bern
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Bern University Hospital, Department of Intensive Care Medicine, Bern University Hospital, and University of Bern, Switzerland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICU Nutr Bern
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2011-03

CONDITIONS: Critical Illness; Starvation; Enteral Nutrition
Keywords: Critical care; Intensive care unit; Early enteral nutrition; Nutritional management protocol
MeSH Terms: conditions — Critical Illness; Starvation | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (Other): Observation
  Interventions: Other: Data Collection
- Nutritional management protocol (Active Comparator): Collection of patient data after implementation of a nutritional management protocol
  Interventions: Other: Nutritional management protocol

INTERVENTIONS:
Other: Data Collection — Collection of patient data before implementation of a nutritional management protocol
  Arms: Observation
Other: Nutritional management protocol — Collection of patient data after implementation of a nutritional management protocol
  Arms: Nutritional management protocol

SUMMARY:
Nutritional treatment has become an essential component of the management of critically ill, due to better knowledge about positive impact of nutritional support. Malnutrition among ICU patients is associated with increased morbidity, mortality, length of stay (LOS) and therefore higher costs.Several studies however suggest, that early implementation of nutritional support is associated with improved clinical outcome, shorter LOS, and decreased infection rates. One of the objectives of this study is to determine if an nutrition protocol can improve the delivery of enteral tube feeding in the ICU.

ELIGIBILITY:
Exclusion Criteria:

* <18 years of age
* stay less than 72 hours on ICU
* die within 72h after admission
* patients admitted for palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Energy delivered (%of caloric target) before and after introducing the nutritional management protocol. | During ICU stay
Protein delivered (% of caloric target) before and after introducing the nutritional management protocol | During ICU stay
Start of enteral feeding after ICU admission | During ICU stay

SECONDARY OUTCOMES:
ICU mortality | During ICU stay
Hospital mortality | During hospital stay
length of ICU stay | During ICU stay
length of hospital stay | During hospital stay
use of antibiotics (days) | During ICU stay
rate of accurately defined infections | During ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Michele Leuenberger, MD, Principal Investigator — University hospital of Bern; Stephan M Jakob, MD, PHD, Study Director — University hospital of Bern; Zeno Stanga, MD, Principal Investigator — University hospital of Bern; Margaret Schafer, MD, Principal Investigator — University hospital of Bern; Jukka Takala, MD, PHD, Study Chair — University hospital of Bern